CLINICAL TRIAL: NCT05353608
Title: Lung Scintigraphy for Pulmonary Embolism Diagnosis in COVID-19 Patients: a Multicenter Observational Study.
Brief Title: Lung Scintigraphy for Pulmonary Embolism Diagnosis in COVID-19 Patients.
Acronym: SCINTI-COVID
Status: Completed | Type: Observational
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: SCINTI-COVID (29BRC21.0143)
Record Dates: First submitted 2022-04-27; First posted 2022-04-29 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2022-04

CONDITIONS: Pulmonary Embolism; COVID-19
Keywords: Lung scintigraphy
MeSH Terms: conditions — Pulmonary Embolism; COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
A frequent complication of COVID-19 disease is pulmonary embolism (PE).

Lung ventilation/perfusion (V/P) scintigraphy is a well-established test for PE diagnosis. The test is interpreted based on the recognition of wedge shaped perfusion mismatched defects. However, the ventilation procedure increases the potential risk of contamination by the aerosol secretion and the expired air.

A variety of strategies have been proposed in the nuclear medicine literature regarding performance of lung ventilation scintigraphy in COVID-19 patients with suspected acute PE. However, there is currently no factual data in this specific population to support recommendations to the nuclear medicine community.

The aim of this study was to assess the role of ventilation imaging when performing lung scintigraphy for suspected PE in COVID-19 patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients with suspected COVID-19 disease
* Referred for lung scintigraphy for suspected acute PE

Exclusion Criteria:

* Patient under guardianship or curatorship
* Patient deprived of liberty by an administrative or judicial decision
* Inability or refuse to give consent

Ages: 18 Years to 99 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: COVID-19 patients who underwent lung scintigraphy for suspected PE.
Sampling Method: Non-Probability Sample
Enrollment: 183 (Actual)
Dates: Start 2021-04-30 (Actual); Primary Completion 2021-05-31 (Actual); Study Completion 2021-05-31 (Actual)

PRIMARY OUTCOMES:
PE diagnosis on lung scintigraphy without the ventilation scan. | 1 day
  Percentage of scans for which the diagnostic conclusion of the lung scan would have been different when omitting the ventilation scan

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - CHRU de Brest, Brest
  - Cnetre Jean-Perrin, Clermont-Ferrand